CLINICAL TRIAL: NCT03286218
Title: A Randomized, Subject- and Investigator-Blind, Placebo and Active-Controlled Study to Assess the Abuse Potential of Lasmiditan
Brief Title: A Study of the Abuse Potential of Lasmiditan in Participants Who Are Recreational Drug Users
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 16853; H8H-MC-LAHB (Other: Eli Lilly and Company)
Record Dates: First submitted 2017-09-15; First posted 2017-09-18 (Actual); Results first posted 2020-01-10 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2017-12

CONDITIONS: Recreational Drug Use; Prescription Drug Abuse (Not Dependent)
MeSH Terms: conditions — Recreational Drug Use; Substance-Related Disorders | interventions — lasmiditan; Alprazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): Placebo was administered orally in one of five treatment periods
  Interventions: Drug: Placebo
- Alprazolam 2 milligram (mg) (Active Comparator): 2 mg of alprazolam was administered orally in one of five treatment periods
  Interventions: Drug: Alprazolam
- Lasmiditan 100 mg (Experimental): 100 mg of lasmiditan was administered orally in one of five treatment periods
  Interventions: Drug: Lasmiditan
- Lasmiditan 200 mg (Experimental): 200 mg of lasmiditan was administered orally in one of five treatment periods
  Interventions: Drug: Lasmiditan
- Lasmiditan 400 mg (Experimental): 400 mg of lasmiditan was administered orally in one of five treatment periods
  Interventions: Drug: Lasmiditan

INTERVENTIONS:
Drug: Lasmiditan — Administered orally
  Other Names: LY573144
  Arms: Lasmiditan 100 mg; Lasmiditan 200 mg; Lasmiditan 400 mg
Drug: Alprazolam — Administered orally
  Arms: Alprazolam 2 milligram (mg)
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the abuse potential of study drug lasmiditan.

Lasmiditan will be compared to a marketed benzodiazepine, alprazolam (positive control), as well as to placebo (dummy substance that looks like lasmiditan or alprazolam without any active drug) to determine the potential for drug abuse. The dosages will be in tablet form and will be taken orally (by mouth).

This study will last about 55 days, including screening. Screening will occur within 28 days prior to qualification phase.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females, as determined by medical history and physical examination.
* Have a body mass index (BMI) of 18 to 32 kilograms per meter squared (kg/m²) inclusive, at the time of screening.
* Must be recreational drug user and agree not to consume any recreational drugs during the study.

Exclusion Criteria:

* Have known allergies to lasmiditan, alprazolam, related compounds, or any components of the formulation, or a history of significant atopy.
* Are currently seeking or participating in treatment for addiction or substance-related disorders, or have recovered from substance abuse disorder.
* Are currently taking excluded prescription or over-the-counter (OTC) medications.
* Have a history of significant sleep disorder, including sleep apnea or narcolepsy.
* Have a history of orthostatic hypotension, vertigo, syncope, or presyncope.
* Have a history of brain injury, including a history of concussions.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2017-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Vince & Associates Clinical Research, Inc., Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Qualification Phase: Participants randomized in a 2-period crossover design with a washout period of at least 72 hours Treatment Phase: Participants randomized to 1 of 10 dosing sequences, irrespective of their qualification randomization, in a 5-period crossover design with a washout period of 3 days in between doses.
Groups:
- Qualification Phase - Alprazolam Then Placebo Sequence 1: Sequence 1 - One tablet of 1 milligram (mg) alprazolam was administered orally in period 1 then placebo period 2.
- Qualification Phase - Placebo Then Alprazolam (Alp) Sequence 2: Sequence 2 - Placebo was administered orally period 1 then one tablet of 2 mg alprazolam period 2.
- Sequence 1: Sequence 1, Periods 1 - 5: (Placebo, 100 mg Las, 2 mg Alp, 200 mg Las, then 400 mg Las)
  All participants received:
  Period 1: Placebo Period 2: 100 mg Las Period 3: 200 mg Las Period 4: 400 mg Las Period 5: 2 mg Alp
  Orally with a 3 day washout between doses.
- Sequence 2: Sequence 2 , Periods 1 - 5: (100 mg Las, 200 mg Las, Placebo, 400 mg Las, then 2 mg Alp)
  All participants received:
  Period 1: 100 mg Las Period 2: 200 mg Las Period 3: Placebo Period 4: 400 mg Las Period 5: 2 mg Alp
  Orally with a 3 day washout between doses.
- Sequence 3: Sequence 3, Periods 1 - 5: (200 mg Las, 400 mg Las, 100 mg Las, 2 mg Alp, then Placebo)
  All participants received:
  Period 1: 200 mg Las Period 2: 400 mg Las Period 3: 100 mg Las Period 4: 2 mg Las Period 5: Placebo
  Orally with a 3 day washout between doses.
- Sequence 4: Sequence 4, Periods 1 - 5: (400 mg Las, 2 mg Alp, 200 mg Las, Placebo, then 100 mg Las)
  All participants received:
  Period 1: 400 mg Las Period 2: 2 mg Alp Period 3: 200 mg Las Period 4: Placebo Period 5: 100 mg Las
  Orally with a 3 day washout between doses.
- Sequence 5: Sequence 5, Periods 1 - 5: (2 mg Alp, Placebo, 400 mg Las, then 200 mg Las)
  All participants received:
  Period 1: 2 mg Alp Period 2: Placebo Period 3: 400 mg Las Period 4: 200 mg Las Period 5: 100 mg Las
  Orally with a 3 day washout between doses.
- Sequence 6: Sequence 6, Periods 1 - 5 (400 mg Las, 200 mg Las, 2 mg Alp, 100 mg Las, then Placebo)
  All participants received:
  Period 1: 400 mg Las Period 2: 200 mg Las Period 3: 2 mg Alp Period 4: 100 mg Las Period 5: Placebo
  Orally with a 3 day washout between doses.
- Sequence 7: Sequence 7, Periods 1-5: (2 mg Alp, 400 mg Las, Placebo, 200 mg Las, then 100 mg Las)
  All participants received:
  Period 1: 2 mg Alp Period 2: 400 mg Las Period 3: Placebo Period 4: 200 mg Las Period 5: 100 mg Las
  Orally with a 3 day washout between doses.
- Sequence 8: Sequence 8, Periods 1 - 5: Placebo, 2 mg Lap, 100 mg Las, 400 mg Las, then 200 mg Las)
  All participants received:
  Period 1: Placebo Period 2: 2 mg Las Period 3: 100 mg Las Period 4: 400 mg Las Period 5: 200 mg Las
  Orally with a 3 day washout between doses.
- Sequence 9: Sequence 9, Periods 1 - 5: (100 mg Las, Placebo, 200 mg Las, 2 mg Alp, 400 mg Las)
  All participants received:
  Period 1: 100 mg Las Period 2: Placebo Period 3: 200 mg Las Period 4: 2 mg Alp Period 5: 400 mg Las
  Orally with a 3 day washout between doses.
- Sequence 10: Sequence 10, Periods 1 - 5: (200 mg Las, 100 mg Las, 400 mg Las, Placebo, then 2 mg Alp)
  All participants received:
  Period 1: 200 mg Las Period 2: 100 mg Las Period 3: 400 mg Las Period 4: Placebo Period 5: 2 mg Alp
  Orally with a 3 day washout between doses.
Period: Qualification Phase Period 1
Arm/Group | Qualification Phase - Alprazolam Then Placebo Sequence 1 | Qualification Phase - Placebo Then Alprazolam (Alp) Sequence 2 | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8 | Sequence 9 | Sequence 10
Started | 48 | 48 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Received at Least One Dose of Study Drug | 47 | 47 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 47 | 47 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Qualification Phase Period 2
Arm/Group | Qualification Phase - Alprazolam Then Placebo Sequence 1 | Qualification Phase - Placebo Then Alprazolam (Alp) Sequence 2 | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8 | Sequence 9 | Sequence 10
Started | 47 | 47 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 30 | 28 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 17 | 19 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Failure to meet randomization criteria | 14 | 15 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Phase Period 1
Arm/Group | Qualification Phase - Alprazolam Then Placebo Sequence 1 | Qualification Phase - Placebo Then Alprazolam (Alp) Sequence 2 | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8 | Sequence 9 | Sequence 10
Started | 0 (Participants completed the Qualification Phase prior to entering the Treatment Phase.) | 0 (Participants completed the Qualification Phase prior to entering the Treatment Phase.) | 6 (Participants completed the Qualification Phase and crossed over to the Treatment Phase.) | 6 (Participants completed the Qualification Phase and crossed over to the Treatment Phase.) | 5 (Participants completed the Qualification Phase and crossed over to the Treatment Phase.) | 6 (Participants completed the Qualification Phase and crossed over to the Treatment Phase.) | 6 (Participants completed the Qualification Phase and crossed over to the Treatment Phase.) | 6 (Participants completed the Qualification Phase and crossed over to the Treatment Phase.) | 6 (Participants completed the Qualification Phase and crossed over to the Treatment Phase.) | 6 (Participants completed the Qualification Phase and crossed over to the Treatment Phase.) | 5 (Participants completed the Qualification Phase and crossed over to the Treatment Phase.) | 6 (Participants completed the Qualification Phase and crossed over to the Treatment Phase.)
Received at Least One Dose of Study Drug | 0 | 0 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 5 | 6
Completed | 0 | 0 | 5 | 5 | 5 | 5 | 6 | 6 | 6 | 6 | 5 | 5
Not Completed | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Period: Treatment Phase Period 2
Arm/Group | Qualification Phase - Alprazolam Then Placebo Sequence 1 | Qualification Phase - Placebo Then Alprazolam (Alp) Sequence 2 | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8 | Sequence 9 | Sequence 10
Started | 0 | 0 | 5 | 5 | 5 | 5 | 6 | 6 | 6 | 6 | 5 | 5
Completed | 0 | 0 | 5 | 5 | 5 | 5 | 6 | 6 | 6 | 6 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Phase Period 3
Arm/Group | Qualification Phase - Alprazolam Then Placebo Sequence 1 | Qualification Phase - Placebo Then Alprazolam (Alp) Sequence 2 | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8 | Sequence 9 | Sequence 10
Started | 0 | 0 | 5 | 5 | 5 | 5 | 6 | 6 | 6 | 6 | 5 | 5
Completed | 0 | 0 | 5 | 5 | 5 | 5 | 6 | 6 | 6 | 6 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Phase Period 4
Arm/Group | Qualification Phase - Alprazolam Then Placebo Sequence 1 | Qualification Phase - Placebo Then Alprazolam (Alp) Sequence 2 | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8 | Sequence 9 | Sequence 10
Started | 0 | 0 | 5 | 5 | 5 | 5 | 6 | 6 | 6 | 6 | 5 | 5
Completed | 0 | 0 | 5 | 5 | 5 | 5 | 6 | 6 | 6 | 6 | 5 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Treatment Phase Period 5
Arm/Group | Qualification Phase - Alprazolam Then Placebo Sequence 1 | Qualification Phase - Placebo Then Alprazolam (Alp) Sequence 2 | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8 | Sequence 9 | Sequence 10
Started | 0 | 0 | 5 | 5 | 5 | 5 | 6 | 6 | 6 | 6 | 5 | 4
Completed | 0 | 0 | 5 | 5 | 5 | 5 | 6 | 6 | 6 | 6 | 5 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Overall Participants: All participants received one dose of alprazolam and placebo in the qualification phase and participants received at least one dose lasmiditan, alprazolam and/or placebo in the treatment phase.
Arm/Group | Overall Participants
Number analyzed (Participants) | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.4 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 91
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 69
  White | 24
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 96

OUTCOME MEASURES:

1. Primary Outcome: Pharmacodynamics (PD): Maximal Effect Score (Emax) of Bipolar Drug Liking Visual Analog Scale (VAS) Scores
Description: The Emax of Bipolar Drug Liking VAS Scores were derived as the maximum at-the-moment Drug Liking VAS score where the time to Emax was the corresponding time point at which the maximum score occurred. The bipolar Drug Liking VAS is consistent with FDA Guidance (January 2017) such that placebo should produce a score between 40 and 60 representing neutral drug-liking (ie, neither like nor dislike); a score ranging from 0 to 100 and a score of 0 indicates strong disliking, and a score of 100 indicates strong liking. Least squares mean (LS mean) was calculated using a linear mixed-effects model, including period, sequence, and treatment as fixed effects, and subject as a random effect, was used to evaluate the hypothesis tests of primary interest (at-the-moment Drug Liking) at the Emax.
Time Frame: Each Phase: 24 Hours
Population: All randomized participants who received at least one dose of study drug had evaluable PD data in each of the 5 periods.
Measure: Least Squares Mean (Standard Error); unit: millimeter (mm)
Groups:
- Alprazolam - 2 mg: 2 mg of Alprazolam administered orally in one of five treatment periods
- Lasmiditan - 100 mg: 100 mg of lasmiditan administered orally in one of five treatment periods
- Lasmiditan - 200 mg: 200 mg of lasmiditan administered orally in one of five treatment periods
- Lasmiditan - 400 mg: 400 mg of lasmiditan administered orally in one of five treatment periods
Arm/Group | Placebo | Alprazolam - 2 mg | Lasmiditan - 100 mg | Lasmiditan - 200 mg | Lasmiditan - 400 mg
Number analyzed (Participants) | 53 | 53 | 53 | 53 | 53
millimeter (mm) | 53.0 (1.94) | 85.4 (1.94) | 68.6 (1.94) | 73.3 (1.94) | 76.6 (1.94)
Statistical Analysis 1: Comparison: Placebo vs Alprazolam - 2 mg; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses versus (vs) Placebo is 14 mm; Least Squares (LS) Mean Difference = 32.4, 90% CI 2-sided [28.4 to 36.4]
Statistical Analysis 2: Comparison: Placebo vs Lasmiditan - 100 mg; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses vs Placebo is 14 mm; LS Mean Difference = 15.6, 90% CI 2-sided [11.7 to 19.6]
Statistical Analysis 3: Comparison: Placebo vs Lasmiditan - 200 mg; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses vs Placebo is 14 mm; LS Mean Difference = 20.3, 90% CI 2-sided [16.3 to 24.3]
Statistical Analysis 4: Comparison: Placebo vs Lasmiditan - 400 mg; Test type: Non-Inferiority — The non-inferiority (NI) margin for Lasmiditan doses vs Placebo is 14 mm; LS Mean Difference = 23.6, 90% CI 2-sided [19.6 to 27.6]
Statistical Analysis 5: Comparison: Alprazolam - 2 mg vs Lasmiditan - 100 mg; Test type: Non-Inferiority — The non-inferiority (NI) margin for Alprazolam and Lasmiditan 100 mg dose is 5 mm; LS Mean Difference = 16.8, 90% CI 2-sided [12.8 to 20.8]
Statistical Analysis 6: Comparison: Alprazolam - 2 mg vs Lasmiditan - 200 mg; Test type: Non-Inferiority — The non-inferiority (NI) margin for Alprazolam and Lasmiditan 200 mg dose is 5 mm; LS Mean Difference = 12.1, 90% CI 2-sided [8.10 to 16.1]
Statistical Analysis 7: Comparison: Alprazolam - 2 mg vs Lasmiditan - 400 mg; Test type: Non-Inferiority — The non-inferiority (NI) margin for Alprazolam and Lasmiditan 400 mg dose is 5 mm; LS Mean Difference = 8.79, 90% CI 2-sided [4.8 to 12.8]

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of Lasmiditan
Description: Pharmacokinetics (PK) defined as the maximum observed drug concentration (Cmax) of lasmiditan
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours Post Dose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Groups:
- Lasmiditan - 200 mg: 200 of lasmiditan administered orally in one of five treatment periods
Arm/Group | Lasmiditan - 100 mg | Lasmiditan - 200 mg | Lasmiditan - 400 mg
Number analyzed (Participants) | 55 | 55 | 55
nanogram/milliliter (ng/mL) | 132 (37) | 299 (35) | 689 (34)

3. Secondary Outcome: PK: Area Under the Curve of Lasmiditan From Zero to Infinity (AUC[0-∞])
Description: PK defined as the area under the curve of lasmiditan from zero to infinity (AUC[0-∞])
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours Post Dose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter (ng*h/mL)
Groups:
- Lasmiditan - 100 mg: 100 mg lasmiditan administered orally in one of five treatment periods
- Lasmiditan - 400 mg Dose: 400 of lasmiditan administered orally in one of five treatment periods
Arm/Group | Lasmiditan - 100 mg | Lasmiditan - 200 mg | Lasmiditan - 400 mg Dose
Number analyzed (Participants) | 55 | 55 | 55
nanogram*hour/milliliter (ng*h/mL) | 856 (32) | 1810 (35) | 3920 (28)

4. Secondary Outcome: PD: Maximal Drug Effects (Emax) Visual Analog Scale (VAS)
Description: Drug Effects VAS Battery lists a series of measures that evaluate different effects of the abuse potential of the study drug. Scales include: Overall drug liking (overall, my liking for this drug is) and ranges from 0 definitely not to 100 definitely so. Take Drug Again (I would take this drug again) and ranges from 0 definitely not to 100 definitely so. Good effects (I can feel good drug effects) and ranges from 0 definitely not to 100 definitely so. Bad effects (I can feel bad drug effects) and ranges from 0 definitely not to 100 definitely so. High (I am feeling) and ranges from 0 not at all high to 100 extremely high. Emax is derived as the maximum score across all postdose time points for each participant. Least Square (LS) Mean is calculated using the linear mixed-effects model with period, sequence and treatment as fixed effects and participant as a random effect.
Time Frame: Each Phase: Predose, 0.25, 0.5, 1, 1.5, 2, 2.5,3, 3.5, 4, 4.5, 5, 6, 8, 12, 24 Hours Post Dose
Population: All randomized participants who received at least one dose of study drug and had evaluable PD data, and completed the study.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Placebo | Alprazolam - 2 mg | Lasmiditan - 100 mg | Lasmiditan - 200 mg | Lasmiditan - 400 mg
Number analyzed (Participants) | 53 | 53 | 53 | 53 | 53
mm
  Overall Drug Liking | 53.1 (2.41) | 86.2 (2.41) | 71.7 (2.41) | 72.2 (2.41) | 77.4 (2.41)
  Take Drug Again | 52.0 (2.70) | 86.0 (2.70) | 71.1 (2.70) | 72.7 (2.70) | 77.3 (2.70)
  Good Effects | 10.8 (4.10) | 80.5 (4.10) | 46.4 (4.10) | 62.9 (4.10) | 63.8 (4.10)
  Bad Effects | 2.47 (3.22) | 22.9 (3.22) | 7.51 (3.22) | 9.75 (3.22) | 15.0 (3.22)
  Any Effects | 8.35 (4.05) | 83.7 (4.05) | 53.3 (4.05) | 65.1 (4.05) | 73.2 (4.04)
  High | 8.61 (3.89) | 77.2 (3.89) | 43.0 (3.89) | 56.1 (3.89) | 67.0 (3.89)
Statistical Analysis 1: Comparison: Placebo vs Alprazolam - 2 mg; Overall Drug Liking; Test type: Other; LS Mean Difference = 33.1, 90% CI 2-sided [28.5 to 37.7]
Statistical Analysis 2: Comparison: Placebo vs Lasmiditan - 100 mg; Overall Drug Liking; Test type: Other; LS Mean Difference = 18.6, 90% CI 2-sided [14.0 to 23.2]
Statistical Analysis 3: Comparison: Placebo vs Lasmiditan - 200 mg; Overall Drug Liking; Test type: Other; LS Mean Difference = 19.1, 90% CI 2-sided [14.5 to 23.8]
Statistical Analysis 4: Comparison: Placebo vs Lasmiditan - 400 mg; Overall Drug Liking; Test type: Other; LS Mean Difference = 24.3, 90% CI 2-sided [19.7 to 28.9]
Statistical Analysis 5: Comparison: Placebo vs Alprazolam - 2 mg; Take drug again; Test type: Other; LS Mean Difference = 34.0, 90% CI 2-sided [29.1 to 38.9]
Statistical Analysis 6: Comparison: Placebo vs Lasmiditan - 100 mg; Take drug again; Test type: Other; LS Mean Difference = 19.1, 90% CI 2-sided [14.2 to 24.0]
Statistical Analysis 7: Comparison: Placebo vs Lasmiditan - 200 mg; Take drug again; Test type: Other; LS Mean Difference = 20.6, 90% CI 2-sided [15.7 to 25.6]
Statistical Analysis 8: Comparison: Placebo vs Lasmiditan - 400 mg; Take drug again; Test type: Other; LS Mean Difference = 25.3, 90% CI 2-sided [20.3 to 30.2]
Statistical Analysis 9: Comparison: Placebo vs Alprazolam - 2 mg; Good effects; Test type: Other; LS Mean Difference = 69.7, 90% CI 2-sided [62.1 to 77.4]
Statistical Analysis 10: Comparison: Placebo vs Lasmiditan - 100 mg; Good effects; Test type: Other; LS Mean Difference = 35.5, 90% CI 2-sided [27.9 to 43.2]
Statistical Analysis 11: Comparison: Placebo vs Lasmiditan - 200 mg; Good effects; Test type: Other; LS Mean Difference = 52.0, 90% CI 2-sided [44.4 to 59.7]
Statistical Analysis 12: Comparison: Placebo vs Lasmiditan - 400 mg; Good effects; Test type: Other; LS Mean Difference = 53.0, 90% CI 2-sided [45.4 to 60.6]
Statistical Analysis 13: Comparison: Placebo vs Alprazolam - 2 mg; Bad effects; Test type: Other; LS Mean Difference = 20.4, 90% CI 2-sided [13.6 to 27.2]
Statistical Analysis 14: Comparison: Placebo vs Lasmiditan - 100 mg; Bad effects; Test type: Other; LS Mean Difference = 5.04, 90% CI 2-sided [-1.76 to 11.8]
Statistical Analysis 15: Comparison: Placebo vs Lasmiditan - 200 mg; Bad effects; Test type: Other; LS Mean Difference = 7.28, 90% CI 2-sided [0.487 to 14.1]
Statistical Analysis 16: Comparison: Placebo vs Lasmiditan - 400 mg; Bad effects; Test type: Other; LS Mean Difference = 12.5, 90% CI 2-sided [5.69 to 19.3]
Statistical Analysis 17: Comparison: Placebo vs Alprazolam - 2 mg; Any effects; Test type: Other; LS Mean Difference = 75.4, 90% CI 2-sided [67.2 to 83.5]
Statistical Analysis 18: Comparison: Placebo vs Lasmiditan - 100 mg; Any effects; Test type: Other; LS Mean Difference = 44.9, 90% CI 2-sided [36.8 to 53.0]
Statistical Analysis 19: Comparison: Placebo vs Lasmiditan - 200 mg; Any effects; Test type: Other; LS Mean Difference = 56.8, 90% CI 2-sided [48.7 to 64.9]
Statistical Analysis 20: Comparison: Placebo vs Lasmiditan - 400 mg; Any effects; Test type: Other; LS Mean Difference = 64.8, 90% CI 2-sided [56.7 to 73.0]
Statistical Analysis 21: Comparison: Placebo vs Alprazolam - 2 mg; High; Test type: Other; LS Mean Difference = 68.6, 90% CI 2-sided [60.6 to 76.6]
Statistical Analysis 22: Comparison: Placebo vs Lasmiditan - 100 mg; High; Test type: Other; LS Mean Difference = 34.4, 90% CI 2-sided [26.4 to 42.4]
Statistical Analysis 23: Comparison: Placebo vs Lasmiditan - 200 mg; High; Test type: Other; LS Mean Difference = 47.5, 90% CI 2-sided [39.5 to 55.5]
Statistical Analysis 24: Comparison: Placebo vs Lasmiditan - 400 mg; High; Test type: Other; LS Mean Difference = 58.4, 90% CI 2-sided [50.4 to 66.3]

5. Secondary Outcome: PD: Maximal Drug Effects (Emax) VAS (Hallucinations)
Description: Drug Effects VAS Battery lists a series of measures that evaluate different effects of the abuse potential of the study drug. The hallucinations scale is presented meaning (I am hallucinating) and ranges from 0 not at all to 100 extremely. Emax is derived as the maximum score across all postdose time points for each participant. Median and interquartile range are reported for each treatment group.
Time Frame: Each Phase: Predose, 0.25, 0.5, 1, 1.5, 2, 2.5,3, 3.5, 4, 4.5, 5, 6, 8, 12, 24 Hours Post Dose
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Placebo | Alprazolam - 2 mg | Lasmiditan - 100 mg | Lasmiditan - 200 mg | Lasmiditan - 400 mg
Number analyzed (Participants) | 53 | 53 | 53 | 53 | 53
mm | 0 [0 to 0] | 0 [0 to 1.00] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Placebo vs Alprazolam - 2 mg; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0
Statistical Analysis 2: Comparison: Placebo vs Lasmiditan - 100 mg; Test type: Superiority; p = 0.0781, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0
Statistical Analysis 3: Comparison: Placebo vs Lasmiditan - 200 mg; Test type: Superiority; p = 0.0625, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0
Statistical Analysis 4: Comparison: Placebo vs Lasmiditan - 400 mg; Test type: Superiority; p = 0.0098, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0

6. Secondary Outcome: PD: Minimum Drug Effects (Emin) Visual Analog Scale (VAS)
Description: Drug Effects VAS Battery lists a series of measures that evaluate different effects of the abuse potential of the study drug. The scales included: Alertness/Drowsiness (I am feeling) ranges from 0 very drowsy to 100 very alert. Agitation/Relaxation (my mood is) and ranges from 0 very relaxed to 100 very agitated. Emin is derived across all postdose time points for each participant. LS Mean was calculated using the linear mixed-effects model with period, sequence and treatment as fixed effects and participant as a random effect.
Time Frame: Each Phase:Predose, 0.25, 0.5, 1, 1.5, 2, 2.5,3, 3.5, 4, 4.5, 5, 6, 8, 12, 24 Hours Post Dose
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Placebo | Alprazolam - 2 mg | Lasmiditan - 100 mg | Lasmiditan - 200 mg | Lasmiditan - 400 mg
Number analyzed (Participants) | 53 | 53 | 53 | 53 | 53
mm
  Alertness/drowsiness | 42.5 (1.97) | 12.5 (1.97) | 25.6 (1.97) | 22.9 (1.97) | 17.7 (1.97)
  Agitation/relaxation | 44.1 (1.94) | 13.4 (1.94) | 24.6 (1.94) | 22.4 (1.94) | 15.4 (1.94)
Statistical Analysis 1: Comparison: Placebo vs Alprazolam - 2 mg; Alertness/drowsiness; Test type: Other; LS Mean Difference = -29.9, 90% CI 2-sided [-34.0 to -25.9]
Statistical Analysis 2: Comparison: Placebo vs Lasmiditan - 100 mg; Alertness/drowsiness; Test type: Other; LS Mean Difference = -16.9, 90% CI 2-sided [-20.9 to -12.8]
Statistical Analysis 3: Comparison: Placebo vs Lasmiditan - 200 mg; Alertness/drowsiness; Test type: Other; LS Mean Difference = -19.6, 90% CI 2-sided [-23.6 to -15.5]
Statistical Analysis 4: Comparison: Placebo vs Lasmiditan - 400 mg; Alertness/drowsiness; Test type: Other; LS Mean Difference = -24.8, 90% CI 2-sided [-28.8 to -20.8]
Statistical Analysis 5: Comparison: Placebo vs Alprazolam - 2 mg; Agitation/relaxation; Test type: Other; LS Mean Difference = -30.8, 90% CI 2-sided [-35.0 to -26.5]
Statistical Analysis 6: Comparison: Placebo vs Lasmiditan - 100 mg; Agitation/relaxation; Test type: Other; LS Mean Difference = -19.5, 90% CI 2-sided [-23.7 to -15.3]
Statistical Analysis 7: Comparison: Placebo vs Lasmiditan - 200 mg; Agitation/relaxation; Test type: Other; LS Mean Difference = -21.7, 90% CI 2-sided [-25.9 to -17.5]
Statistical Analysis 8: Comparison: Placebo vs Lasmiditan - 400 mg; Agitation/relaxation; Test type: Other; LS Mean Difference = -28.8, 90% CI 2-sided [-33.0 to -24.5]

7. Secondary Outcome: PD: Mean Scores on Drug Similarity VAS Measures
Description: Participants marked a point on a 100-mm horizontal line that best represented their response to the given question. The endpoints of each electronic scale were marked with descriptive anchors on a scale from 0 to 100 (Fraser et al. 1961; Bond and Lader 1974; Bigelow 1991; Shram et al. 2010). In the "How similar" questions, ranges from 0 to 100 and a score of 0 indicates definitely not similar, and a score of 100 indicates definitely similar.
Time Frame: Each Phase: 24 Hours Post Dose
Population: All randomized participants who received at least one dose of study drug, were familiar with each listed drug on the questionnaire and had evaluable data.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo - Qualification Phase: Placebo was administered orally in one of 2 treatment periods.
- 1 mg Alprazolam - Qualification Phase: 1 mg of Alprazolam was administered orally in one of 2 treatment periods.
- 2 mg Alprazolam: 2 mg of Alprazolam was administered orally in one of five treatment periods.
Arm/Group | Placebo - Qualification Phase | 1 mg Alprazolam - Qualification Phase | Placebo | 2 mg Alprazolam | Lasmiditan - 100 mg | Lasmiditan - 200 mg | Lasmiditan - 400 mg
Number analyzed (Participants) | 95 | 94 | 55 | 53 | 55 | 55 | 55
score on a scale
  How similar with cocaine /: number analyzed (Participants) | 50 | 51 | 28 | 27 | 28 | 28 | 27
  How similar with cocaine / | 1.3 (3.5) | 5.8 (10.6) | 2.2 (6.6) | 6.1 (13.6) | 2.7 (4.2) | 14.6 (26.3) | 12.5 (23.3)
  How similar with caffeine: number analyzed (Participants) | 74 | 73 | 43 | 42 | 44 | 44 | 43
  How similar with caffeine | 2.9 (10.3) | 3.2 (6.0) | 1.5 (7.2) | 4.4 (9.7) | 2.2 (2.4) | 4.4 (9.8) | 4.1 (8.3)
  How similar to MDMA (Ectasy): number analyzed (Participants) | 31 | 31 | 18 | 17 | 17 | 18 | 17
  How similar to MDMA (Ectasy) | 4.7 (13.5) | 10.0 (20.4) | 1.4 (3.9) | 20.5 (23.7) | 10.6 (19.9) | 17.1 (28.2) | 18.7 (28.2)
  How similar to amphetamine or methamphetamine: number analyzed (Participants) | 24 | 24 | 16 | 15 | 16 | 17 | 16
  How similar to amphetamine or methamphetamine | 1.5 (5.4) | 4.3 (6.3) | 2.4 (6.0) | 3.9 (5.5) | 2.3 (2.5) | 4.6 (4.8) | 4.4 (6.2)
  How similar to phencyclidine (PCP): number analyzed (Participants) | 3 | 4 | 3 | 3 | 3 | 3 | 3
  How similar to phencyclidine (PCP) | 22.0 (30.6) | 0.5 (1.0) | 0.0 (0.0) | 26.7 (40.3) | 1.3 (1.5) | 24.0 (37.3) | 32.3 (43.7)
  How similar to codeine or morphine use: number analyzed (Participants) | 83 | 82 | 49 | 47 | 49 | 49 | 49
  How similar to codeine or morphine use | 11.4 (23.8) | 41.5 (35.1) | 8.1 (21.7) | 50.8 (31.2) | 30.9 (30.4) | 37.6 (31.7) | 45.9 (32.4)
  How similar to (lysergic acid diethylamide (LSD): number analyzed (Participants) | 11 | 12 | 6 | 6 | 6 | 7 | 6
  How similar to (lysergic acid diethylamide (LSD) | 1.2 (3.9) | 4.1 (6.9) | 4.2 (6.6) | 6.2 (7.5) | 3.5 (4.6) | 5.9 (5.5) | 7.2 (8.0)
  How similar to nicotine: number analyzed (Participants) | 77 | 76 | 44 | 42 | 44 | 43 | 44
  How similar to nicotine | 2.9 (11.8) | 5.1 (9.6) | 1.4 (5.5) | 3.8 (9.4) | 3.3 (11.0) | 3.6 (9.0) | 4.3 (8.6)
  How similar to cannabis: number analyzed (Participants) | 92 | 91 | 53 | 51 | 53 | 53 | 53
  How similar to cannabis | 10.8 (24.7) | 39.9 (33.5) | 8.9 (22.9) | 51.2 (30.3) | 29.9 (30.0) | 37.4 (29.6) | 41.7 (31.6)
  How similar to benzodiazepine: number analyzed (Participants) | 94 | 93 | 55 | 53 | 55 | 55 | 55
  How similar to benzodiazepine | 14.4 (32.4) | 75.9 (36.2) | 13.1 (30.6) | 88.1 (22.6) | 57.2 (40.3) | 66.9 (38.7) | 74.6 (31.9)
  How similar to mushrooms: number analyzed (Participants) | 14 | 15 | 7 | 7 | 7 | 8 | 7
  How similar to mushrooms | 0.0 (0.0) | 2.7 (3.8) | 2.1 (5.2) | 3.7 (6.1) | 2.1 (2.1) | 3.8 (5.7) | 4.9 (6.3)
  How similar to heroin: number analyzed (Participants) | 4 | 5 | 2 | 2 | 2 | 2 | 2
  How similar to heroin | 0.0 (0.0) | 17.8 (38.1) | NA (NA) — Mean and standard deviation are not calculated due to N=2, minimum and maximum values are reported: minimum value is 0 and maximum value is 0. | NA (NA) — Mean and standard deviation are not calculated due to N=2, minimum and maximum values are reported: minimum value is 0 and maximum value is 79. | NA (NA) — Mean and standard deviation are not calculated due to N=2, minimum and maximum values are reported: minimum value is 0 and maximum value is 3. | NA (NA) — Mean and standard deviation are not calculated due to N=2, minimum and maximum values are reported: minimum value is 2 and maximum value is 60. | NA (NA) — Mean and standard deviation are not calculated due to N=2, minimum and maximum values are reported: minimum value is 2 and maximum value is 96.

ADVERSE EVENTS:
Time Frame: From Baseline to Study Completion (Up to 2 months)
Description: All randomized participants who received at least one dose of study drug.
Groups:
- Qualification Phase - Placebo: Placebo was administered orally.
- Qualification Phase - Alprazolam: 1 mg of alprazolam was administered orally.
- Treatment Phase - Placebo: Placebo was administered orally in one of five treatment periods.
- Treatment Phase - 2 mg Alprazolam: 2 mg alprazolam was administered orally in one of five treatment periods.
- Treatment Phase - 100 mg Lasmiditan: 100 mg of Lasmiditan was administered orally in one of five treatment periods.
- Treatment Phase - 200 mg Lasmiditan: 200 mg of Lasmiditan was administered orally in one of five treatment periods.
- Treatment Phase - 400 mg Lasmiditan: 400 mg of Lasmiditan was administered orally in one of five treatment periods.
Arm/Group | Qualification Phase - Placebo | Qualification Phase - Alprazolam | Treatment Phase - Placebo | Treatment Phase - 2 mg Alprazolam | Treatment Phase - 100 mg Lasmiditan | Treatment Phase - 200 mg Lasmiditan | Treatment Phase - 400 mg Lasmiditan
All-Cause Mortality (participants affected / at risk) | 0/95 | 0/94 | 0/55 | 0/53 | 0/55 | 0/55 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/95 | 0/94 | 0/55 | 0/53 | 0/55 | 0/55 | 0/55
Other Adverse Events (participants affected / at risk) | 8/95 | 74/94 | 12/55 | 49/53 | 33/55 | 42/55 | 47/55
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Qualification Phase - Placebo (N=95) | Qualification Phase - Alprazolam (N=94) | Treatment Phase - Placebo (N=55) | Treatment Phase - 2 mg Alprazolam (N=53) | Treatment Phase - 100 mg Lasmiditan (N=55) | Treatment Phase - 200 mg Lasmiditan (N=55) | Treatment Phase - 400 mg Lasmiditan (N=55)
Feeling of relaxation (General disorders) | 3 (3) | 20 (20) | 1 (1) | 12 (12) | 6 (6) | 4 (4) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 10 (10) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 6 (6) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 4 (5) | 4 (4) | 3 (4) | 3 (3) | 4 (4)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 6 (6) | 5 (5)
Somnolence (Nervous system disorders) | 3 (3) | 52 (52) | 2 (2) | 45 (45) | 18 (18) | 22 (22) | 30 (30)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 3 (3) | 2 (2)
Euphoric mood (Psychiatric disorders) | 1 (1) | 22 (22) | 6 (6) | 23 (23) | 14 (14) | 27 (27) | 25 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-09-05): https://cdn.clinicaltrials.gov/large-docs/18/NCT03286218/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-11): https://cdn.clinicaltrials.gov/large-docs/18/NCT03286218/SAP_001.pdf